CLINICAL TRIAL: NCT01526512
Title: Low Dose of Metronomic Cyclophosphamide and Capecitabine in Pretreated HER2-negative Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, yanfei Liu, Principal investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: metroCX
Record Dates: First submitted 2012-01-29; First posted 2012-02-06 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Metronomic cyclophosphamide; Metronomic capecitabine; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metroCX (Experimental): metroCX Cyclophosphamide 50mg PO d1-28; Capecitabine 1500mg PO d1-28; every 28days
  Interventions: Drug: metroCX

INTERVENTIONS:
Drug: metroCX — cyclophosphamide 50mg PO d1-28 capecitabine 1500mg PO d1-28; every 28days

SUMMARY:
The purpose of this study is to evaluate the role of low dose metronomic cyclophosphamide and capecitabine in pretreated metastatic breast cancer.

DETAILED DESCRIPTION:
Metronomic chemotherapy has been considered as an effective strategy in metastatic breast cancer. This trial is designed to evaluate the role of low dose metronomic cyclophosphamide and capecitabine in pretreated metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 80 years old
2. ECOG performance between 0-3
3. Life expectancy more than 3 months
4. Histological proven unresectable recurrent or advanced HER2-negative breast cancer
5. At least one previous therapy regimen (including endocrine therapy) for metastatic breast cancer;suitable for monotherapy (Neoadjuvant or adjuvant docetaxel should be completed at least one year).
6. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST1.1)
7. No anticancer therapy within 4 weeks
8. Adequate hematologic, hepatic, and renal function,No serious medical history of heart, lung, liver and kidney
9. Provision of written informed consent prior to any study specific procedures
10. Previous capecitabine is permitted, however, it should be completed at least 6 months.

Exclusion Criteria:

1. Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound)
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the course of the study
3. Treatment with an investigational product within 4 weeks before the first treatment
4. Symptomatic central nervous system metastases
5. Other active malignancies (including other hematologic malignancies) or other malignancies, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
6. Patient having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
7. Uncontrolled serious infection
8. Patients with bad compliance
9. Patients lack of Dihydropyrimidine Dehydrogenase(DPD)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks

SECONDARY OUTCOMES:
Biomarker | 6 weeks
  Relationship of serum VEGF level and efficacy
Biomarker | 6weeks
  Relationship of immuno-marker(CD3,CD4,CD8,etc) and efficacy
Biomarker | 1 time
  Relationship of genetics(genetic polymorphisms) and efficacy
Efficacy | 6 weeks
  Overall Response rate
Efficacy | 6 weeks
  Overall Survival
Safety | 3 weeks
  Safety（NCI CTCAE v4.0）

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China